CLINICAL TRIAL: NCT05705453
Title: Epidural Stimulation After Neurologic Damage: Long-Term Outcomes
Acronym: LTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2022-365
Record Dates: First submitted 2023-01-04; First posted 2023-01-30 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: SCI - Spinal Cord Injury
Keywords: spinal cord stimulation; epidural stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Volitional EMG power (Experimental): Assessing the change in volitional EMG power during the Brain Motor Control Assement (BMCA) between nonstimulation baseline and stimulation.
  Interventions: Device: Epidural Spinal Cord Stimulation

INTERVENTIONS:
Device: Epidural Spinal Cord Stimulation — Stimulation of the spinal cord from the epidural space.

SUMMARY:
This study will evaluate the long-term effect of chronic spinal cord stimulation to restore volitional movement for patients with chronic spinal cord injuries.

DETAILED DESCRIPTION:
Participants will be enrolled in this study for the duration of 10 years. They will need to come to Minneapolis twice a year for the Brain Motor Control Assessment and will be given different settings within their Spinal Cord Stimulator (SCS) programing.

ELIGIBILITY:
Inclusion Criteria:

* 22 years of age or older
* Able to undergo the informed consent process
* Stable spinal cord injury
* International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) neurologic level of injury below C5
* No ventilator dependency within the last year
* American Spinal Injury Association (AISA) imparement scale"A" or "B" in the absence of spinal cord stimulation
* Medically stable in the judgment of the Principal investigator
* Greater than 1 year since initial injury and at least 6 months from any required spinal instrumentation and 2 months from spinal cord stimulator surgery
* Has an existing and functional implanted spinal cord stimulator system that is FDA approved and can be corroborated by hospital documentation
* Spinal imaging of the stimulator system

Exclusion Criteria:

* Current and anticipated need for opioid pain medications or pain that would prevent full participation in the rehabilitation program in the judgment of the principal investigator
* Use of botulinum toxin (Botox) injections in the previous six months
* Clinically significant mental illness in the judgment of the principal investigator
* Other conditions or medications that would make the subject unable to participate in testing/rehabilitation in the judgment of the principal investigator
* Nonfunctional spinal cord stimulator or near end-of-life, determined by the PI
* Current Pregnancy
* Current pain relief from the spinal cord stimulator if the indication for implantation was for management of chronic pain.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2033-04-01 (Estimated); Study Completion 2034-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Volitional electromyography (EMG) power | 10 years
  The measurement of volitional change using EMG during the Brain Motor Control assessment between nonstimulation baseline and stimulation

SECONDARY OUTCOMES:
Prediction of power preferences | 10 years
  Prediction of power of preference models built based on evaluations of stimulation settings.

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, MD, Principal Investigator — University of Minnesota
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trial Website — http://estand.org